CLINICAL TRIAL: NCT02142660
Title: Prospective Study Evaluating the Usefulness of Sprayshield as Adhesion Barrier System in Two Steps Laparoscopic Bariatric Surgery for Obese Patients
Brief Title: Sprayshield as Adhesion Barrier System for Obese Patients
Acronym: Sprayshield
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: UF8744
Record Dates: First submitted 2012-03-05; First posted 2014-05-20 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-04

CONDITIONS: Severe Obesity
Keywords: Adhesion barrier system; Bariatric surgery
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sprayshield: Applied to the operating zone during an ablation of gastric died ring at obese patients programmed for the second bariatric surgery to type of bypass gastric or of gastrectomie
  Interventions: Procedure: ablation of gastric

INTERVENTIONS:
Procedure: ablation of gastric — Applied to the operating zone during an ablation of gastric died ring at obese patients programmed for the second bariatric surgery to type of bypass gastric or of gastrectomie in wing

SUMMARY:
The application of SprayShield during a laparoscopic band removal (first surgical step) will be evaluated to see if the postoperative adhesions between the stomach, the left liver and the diaphragm are not severe, facilitating the surgical surgical step of a gastric bypass or a sleeve gastrectomy.

DETAILED DESCRIPTION:
Monocenter and observational study on 20 obese patients, requiring removal of the gastric band for poor results (weight regain or insufficient weight-loss) or mechanical complications of the band ( slippage, esophageal dilation) and schedule for a second step surgery of gastric bypass or sleeve gastrectomy 2 months later.

ELIGIBILITY:
Inclusion Criteria:

* Obese male or female who would benefit from a gastric band removal and for whom a second surgical step with conversion to sleeve gastrectomy or bypass is scheduled

Exclusion Criteria:

* The patients having an ablation of ring motivated for an infectious complication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese male or female who would benefit from a gastric band removal and for whom a second surgical step with conversion to sleeve gastrectomy or bypass is scheduled
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
During the second surgical step the intensity of the adhesions in the operative field will be determined by the adhesion surface area and the adhesion intensity using | intra operative
  During Conversion in Bypass or Sleeve Gastrectomy the intensity of the adhesions in the operative field will be determined by the adhesion surface area and the adhesion intensity using a 4-point : scale 0 (no adhesion), 1 (fine and esily detachable adhesions), 2 (thick vascularize adhesion), 3 (intense adhesion preventing the identification of cleavable plane between organs)

SECONDARY OUTCOMES:
Duration of surgery | 30 day surgical mortility
  Duration of surgery 30 day surgical mortility

CONTACTS AND LOCATIONS:
Overall Officials: Jean Michel FABRE, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Department of Digestive Surgery A, Saint Eloi Hospital, Montpellier, France

REFERENCES:
- [Result] Nocca D, Guillaume F, Noel P, Picot MC, Aggarwal R, El Kamel M, Schaub R, de Seguin de Hons C, Renard E, Fabre JM. Impact of laparoscopic sleeve gastrectomy and laparoscopic gastric bypass on HbA1c blood level and pharmacological treatment of type 2 diabetes mellitus in severe or morbidly obese patients. Results of a multicenter prospective study at 1 year. Obes Surg. 2011 Jun;21(6):738-43. doi: 10.1007/s11695-011-0385-2. PMID 21468625
- [Result] Fezzi M, Kolotkin RL, Nedelcu M, Jaussent A, Schaub R, Chauvet MA, Cassafieres C, Lefebvre P, Renard E, Bringer J, Fabre JM, Nocca D. Improvement in quality of life after laparoscopic sleeve gastrectomy. Obes Surg. 2011 Aug;21(8):1161-7. doi: 10.1007/s11695-011-0361-x. PMID 21298508
- [Result] Blanc PM, Lagoutte JM, Picot MC, Deneve E, de Seguin C, Fabre JM, Nocca D. Preliminary results of the laparoscopic adjustable gastric banding procedure by a new generation of silicone band: MIDBAND. Obes Surg. 2008 May;18(5):569-72. doi: 10.1007/s11695-008-9441-y. PMID 18340499
- [Result] Nocca D, Krawczykowsky D, Bomans B, Noel P, Picot MC, Blanc PM, de Seguin de Hons C, Millat B, Gagner M, Monnier L, Fabre JM. A prospective multicenter study of 163 sleeve gastrectomies: results at 1 and 2 years. Obes Surg. 2008 May;18(5):560-5. doi: 10.1007/s11695-007-9288-7. PMID 18317859
- [Result] Nocca D, Aggarwal R, Blanc P, Gallix B, Di Mauro GL, Millat B, Seguin des De Hons C, Deneve E, Rodier JG, Tincani G, Pierredon MA, Fabre JM. Laparoscopic vertical banded gastroplasty. A multicenter prospective study of 200 procedures. Surg Endosc. 2007 Jun;21(6):870-4. doi: 10.1007/s00464-006-9048-0. Epub 2006 Nov 14. PMID 17103270